CLINICAL TRIAL: NCT07057635
Title: Wireless Irradiance SEnsors During Neonatal Phototherapy: The WISE Clinical Study
Brief Title: Wireless Irradiance SEnsors During Neonatal Phototherapy
Acronym: WISE
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Guilherme Sant'Anna, MD, Neonatologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: WISE Clinical
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Hyperbilirubinemia; Jaundice, Neonatal; Phototherapy Complication; Newborn Complication
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Extremely Preterm Infant: Weighing < 1500g at recruitment.
- Late Preterm Infant: Weighing between between 1500g and 2500g at recruitment.
- Term Infant: Weighing > 2500g at recruitment.

SUMMARY:
Bilisensors are devices designed to measure the cumulative dose of phototherapy administered to neonates undergoing treatment for hyperbilirubinemia. The current standard of care typically involves intermittent spot measurements once a day using a handheld dosimeter that may give variable estimations. In contrast, bilisensors may enable continuous, real-time monitoring of light exposure, helping to know the total phototherapy dose received by the infant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be admitted to the Montreal Children's Hospital (MCH) Neonatal Intensive Care Unit (NICU)
* Under phototherapy as clinically indicated
* Diagnosis of indirect hyperbilirubinemia
* Weight of >1000g at time of enrollment

Exclusion Criteria:

* Any abnormal skin conditions (example: extreme dryness, desquamation, congenital skin disorders, etc.)
* Diagnosis of direct hyperbilirubinemia
* Weight of <1000g at time of enrollment
* Any baby or family deemed ineligible (ex. too much stress, too unstable) by the clinical care team

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any micro premature, preterm or term neonate admitted to NICU undergoing phototherapy due to indirect hyperbilirubinemia will be considered for this pilot study. A convenience sample size of 6 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Light Intensity | 3 Hours
  Comparison of intensity (µW/cm^2) data between the Wearifi Bili Light Dosimeter and gold-standard Ohmeda BiliBlanket Light meter at 3 time points: start, 1.5 h and end.

SECONDARY OUTCOMES:
Cumulative Dose | 3 Hours
  To determine the cumulative phototherapy dose (µ J/cm^2) measured with the Wearifi Bili Light Dosimeter during the study period.
Data Transmission & Gaps | 2 Months
  Evaluation of data transmission and possible gaps from the Wearifi Bili Light Dosimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Sant'Anna, MD, PhD, Principal Investigator — RI-MUHC

IPD SHARING:
Plan to Share IPD: No